CLINICAL TRIAL: NCT01569516
Title: A Phase II, Double Blind, Placebo-controlled, Randomized, Multi-Center, Parallel Group Dose Exploring Study to Evaluate the Efficacy and Safety of Octohydroaminoacridine Succinate Tablets in Patient With Mild to Moderate Alzheimer's Disease
Brief Title: Study of Octohydroaminoacridine Succinate Tablets in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun Huayang High-tech Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCHY2010L00161-HPAD2
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2011-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Octohydroaminoacridine Succinate
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low dose (Experimental): 1mg, tid
  Interventions: Drug: Octohydroaminoacridine Succinate Tablets
- Moderate dose (Experimental): 2mg,tid
  Interventions: Drug: Octohydroaminoacridine Succinate Tablets
- High dose (Experimental): 4mg,tid
  Interventions: Drug: Octohydroaminoacridine succinate Tablets
- Placebo (Placebo Comparator): 0 mg, tid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octohydroaminoacridine Succinate Tablets — 1mg, tid
  Arms: low dose
Drug: Octohydroaminoacridine Succinate Tablets — 1st-2nd week, 1mg, tid 3rd -16th week, 2mg, tid
  Arms: Moderate dose
Drug: Octohydroaminoacridine succinate Tablets — 1st-2nd week, 1mg, tid, 3rd -4th week, 2mg, tid, 5th-16th week, 4mg, tid
  Arms: High dose
Drug: Placebo — 0mg, tid
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of Octohydroaminoacridine Succinate tablets and find the optimal dose in patients with mild to moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
The purpose of this study is a preliminary assessment of the Octohydroaminoacridine Succinate tablets in the treatment of mild to moderate Alzheimer's disease and explore the efficacy and safety of the best dose. The 288 patients were randomly assigned to four groups: high dose (4mg / time), moderate dose (2mg / time), low dose (1mg / time) and the placebo group, including four weeks of the trial screening period following 16 weeks double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of probable AD based on DSM-IV and the NINCDS-ADRDA criteria.
2. Male/female patient aged between 50 and 85.
3. mild to moderate probable AD ：Middle school or above: 11 ≤MMSE ≤ 25, elementary school: 8 ≤ MMSE ≤ 20, illiteracy: 5 ≤ MMSE ≤ 16.
4. CT or MRI scan excluding another structural brain disease in one year.
5. Neurologic examination no significant abnormalities.
6. Hachinski Ischemic Score < 4；Hamilton Depression Scale ≤10. Able to complete the test procedure, audio-visual and physical ability to act to complete the neuropsychological measure.
7. Stable chaperone, more than 2 hours a day together with the patient or accumulated fewer than 14 hours per week.
8. Informed consent of the patient (or legal representative) and of the caregiver agreeing to take part in the study.

Exclusion Criteria:

1. Proven or clinically suspected other type of dementia such as vascular dementia, Lewy body dementia, Parkinson's disease, frontotemporal dementia, g - Jakob disease (spastic pseudo-sclerosis), normal pressure hydrocephalus etc.
2. Sudden onset of early dementia or with gait disorders, seizures and behavioral changes.
3. Clinical manifestations of focal neurological signs (hemiparesis, sensory loss, visual field defect) or early extrapyramidal tract signs.
4. History of cerebrovascular disease and stroke.
5. Serious lack of folic acid and VitB12, syphilis antibody positive or thyroid dysfunction.
6. Mechanical intestinal obstruction patient ,Resting pulse less than 60,Severe liver or renal disease.
7. Patients with mechanical intestinal obstruction.
8. History of bone marrow transplantation.Mental illness, such as severe depression.
9. Cognitive damage caused by alcohol or drug abuse. Disable to correctly evaluate the cognitive function.
10. Critical condition, disable to make the exact evaluation of the efficacy and safety of new drug.
11. Use of any agent for the treatment of dementia within 4 weeks of randomization.
12. Be sensitive to ACHEI.
13. Be sensitive to two or more foods/drugs.
14. Use of another investigational agent within one months of screening.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale | 20weeks

SECONDARY OUTCOMES:
Clinician's Interview Based Impression of Change, plus caregiver input | 20weeks
Activities of Daily Living:Activities of Daily Living Scale（ADL) | 20weeks
Mental behavior: neuropsychiatric questionnaire (NPI) | 20weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shifu Xiao, MD, Principal Investigator — Shanghai Mental Health Center
Locations (13):
- China (13):
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Hebei mental health center, Baoding, Hebei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first Affiliated Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Beijing HuiLongGuan Hospital, Beijing
  - Beijing Shijitan Hospital, EMU, Beijing
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Tenth People's hospital, Shanghai
  - Shanghai, Shanghai